CLINICAL TRIAL: NCT02462343
Title: Comparison of the Two and Six- Minute Walk Tests in Evaluating Oxygen Desaturation in Patients With Severe COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Schön Klinik Berchtesgadener Land (Other)
Responsible Party: Principal Investigator, Klaus Kenn, MD, Schön Klinik Berchtesgadener Land
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: walk test trial
Record Dates: First submitted 2015-06-02; First posted 2015-06-04 (Estimated); Last update posted 2015-06-04 (Estimated); Status verified 2015-06

CONDITIONS: Chronic Obstructive Lung Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 minute walk test (Other)
  Interventions: Other: walk tests
- 6 minute walk test (Other)
  Interventions: Other: walk tests

INTERVENTIONS:
Other: walk tests

SUMMARY:
All measurements are performed on two consecutive days at the beginning of a pulmonary rehabilitation program in a randomized cross-over study design. On the first day, each patient is randomly assigned to perform either the 2 minute walk test or the 6 Minute walk test. On the second day each patient performs the test that was not performed on the first day. All walk tests are performed by the same investigator on the same track and time of day, following the 2002 guidelines of the American Thoracic Society.

Patients wear a mobile pulse oximeter that continuously records heart rate and oxygen saturation during testing. Baseline values of oxygen saturation, heart rate and ratings of perceived exertion on the modified Borg scale (0 to 10) for dyspnea and leg fatigue are recorded at rest after 10 minutes of sitting.

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis of chronic obstructive lung disease stage III or IV according to the Global Initiative for chronic Obstructive Lung Diseases definition
* ability to read and understand the German language and study procedures.
* written informed consent

Exclusion Criteria:

* severe acute exacerbation of chronic obstructive lung disease
* severe respiratory failure (partial Oxygen pressure at rest lower than 55 millimeter mercury)
* non compliance to the study protocol.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2007-03; Primary Completion 2007-05 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
oxygen desaturation | up to 6 minute walk test

SECONDARY OUTCOMES:
heart rate | during 2 minute walk test and 6 minute walk test
perceived exertion for dyspnea and leg fatigue | during 2 minute walk test and 6 minute walk test
  measured by a modified Borg scale from 0 to 10

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Kenn, MD, Principal Investigator — Schoen Klinik Berchtesgadener Land